CLINICAL TRIAL: NCT03112291
Title: Clinical and Microbiological Evaluation of a Series of Clinical Cases of Permanent Teeth With Incomplete Apexogenesis and Traumatic Necrosis, Treated With Double Antimicrobial Paste, Revascularization Procedures, and MTA
Brief Title: Antimicrobial Pastes and Clinical Cases of Apexogenesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adriana Kelly de Sousa Santiago Barbosa (Other)
Responsible Party: Sponsor-Investigator, Adriana Kelly de Sousa Santiago Barbosa, PhD, Universidade Federal do Ceara
Organization: Universidade Federal do Ceara (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Estudo Clinico - Apicificação
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Apexification; Root Canal Therapy; Dental Trauma
Keywords: anti-microbial agents; apexification; dental pulp; endodontics; root canal therapy; dental trauma
MeSH Terms: interventions — Apexification

STUDY DESIGN:
Intervention Model Description: This investigation is a longitudinal prospective interventional study of a series of cases
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- permanent teeth apexification (Experimental): They should have one permanent tooth with traumatic necrosis, which in turns should show color alteration, fistulae, periapical lesion, and/or internal or external root resorption, pain, or absence of pulp response to sensitivity tests at a clinical examination to be considered necrotic. Male and female patients who had not undergone antibiotic therapy 3 months before the treatment were included and clinical and radiographic examinations confirmed pulp necrosis. This study analyzed the clinical and microbiological results of the endodontic treatment performed on permanent teeth with necrosis caused by traumatic injury and treated using revascularization technique, double antibiotic paste, intra-canal medication, and an MTA cervical plug.
  Interventions: Procedure: Apexification

INTERVENTIONS:
Procedure: Apexification — Apexification forms a calcified barrier in teeth with open apexes and pulp necrosis. It is used to treat immature teeth, but it does not promote the continuity of root formation.
  Other Names: Pulp Revascularization

SUMMARY:
The aim of this study was to perform a clinical and microbiological evaluation of teeth with incomplete apexogenesis and traumatic necrosis that were treated with a revascularization technique, evaluating the microbial reduction after the use a double antibiotic paste. Furthermore, the investigation also aims to identify the presence of Enterococcus faecalis and Porphyromomas gingivalis within the root canal system.

DETAILED DESCRIPTION:
This investigation is a longitudinal prospective interventional study of a series of cases. Patients who sought treatment at the Faculty of Dentistry from June 2011 to September 2015 were selected. They should have one permanent tooth with traumatic necrosis.

ELIGIBILITY:
Inclusion Criteria:

* They should have one permanent tooth with traumatic necrosis, which in turns should show color alteration, fistulae, periapical lesion, and/or internal or external root resorption, pain, or absence of pulp response to sensitivity tests at a clinical examination to be considered necrotic. Male and female patients who had not undergone antibiotic therapy 3 months before the treatment were included and clinical and radiographic examinations confirmed pulp necrosis.

Exclusion Criteria:

* Patients who did use antibiotics
* Patients who did loss of temporary coronary sealing between treatment sessions
* Patients who give up the research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-11-25 (Actual); Primary Completion 2015-06-10 (Actual); Study Completion 2016-10-08 (Actual)

PRIMARY OUTCOMES:
Number of teeth with apex closed according to nolle stages. | 24 months
  The apical closure of the teeth was evaluated by radiography /computed tomography every 3 months according to the nolla stages, in which a tooth is considered to be a closed apex in stage 9 of nolla

SECONDARY OUTCOMES:
Number of patients with clinically and radiographically observed fistulas | 6 months
  The occurrence of fistulas through clinical signs and symptoms was observed for a period of 6 months in which it was recorded in medical records

CONTACTS AND LOCATIONS:
Overall Officials: José Jeová S Moreira Neto, Dr, Study Director — Universidade Federal do Ceará
Locations (1):
- Adriana Kelly de Sousa Santiago Barbosa, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pace R, Giuliani V, Nieri M, Di Nasso L, Pagavino G. Mineral trioxide aggregate as apical plug in teeth with necrotic pulp and immature apices: a 10-year case series. J Endod. 2014 Aug;40(8):1250-4. doi: 10.1016/j.joen.2013.12.007. Epub 2014 Apr 3. PMID 25069943
- [Result] Nagata JY, Gomes BP, Rocha Lima TF, Murakami LS, de Faria DE, Campos GR, de Souza-Filho FJ, Soares Ade J. Traumatized immature teeth treated with 2 protocols of pulp revascularization. J Endod. 2014 May;40(5):606-12. doi: 10.1016/j.joen.2014.01.032. Epub 2014 Mar 6. PMID 24767551
- [Result] Trope M. Treatment of the immature tooth with a non-vital pulp and apical periodontitis. Dent Clin North Am. 2010 Apr;54(2):313-24. doi: 10.1016/j.cden.2009.12.006. PMID 20433980